CLINICAL TRIAL: NCT00729716
Title: Phase II Study to Investigate the Efficacy and Safety of BioCart™II in the Treatment of Symptomatic Cartilage Defects of the Femoral Condyle in Comparison With Microfracture
Brief Title: Comparison of BioCart™II With Microfracture for Treatment of Cartilage Defects of the Femoral Condyle
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ProChon Biotech Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BioCart™II 005-06
Record Dates: First submitted 2008-08-04; First posted 2008-08-07 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-03

CONDITIONS: Symptomatic Cartilage Defects of the Femoral Condyle
Keywords: Microfracture; Cartilage repair; Autologous chondrocyte implantation
MeSH Terms: conditions — Fractures, Stress | interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): BioCart™II treatment
  Interventions: Biological: BioCart™II
- B (Active Comparator): Microfracture procedure
  Interventions: Procedure: Microfracture

INTERVENTIONS:
Biological: BioCart™II — A cartilage biopsy will be harvested from patients during arthroscopy and used for chondrocyte isolation, culture and future implantation. Subjects will also have about 80 ml venous blood drawn for autologous cell culture medium. Two-four weeks following biopsy harvest, BioCart™II will be implanted into the cartilage defect after careful debridement via miniarthrotomy.
  Other Names: Autologous chondrocyte implantation; ACI
  Arms: A
Procedure: Microfracture — MF procedure will be carried out according to accepted practice. After careful debridement multiple perforations, or microfractures, are made in the subchondral bone using an awl. The released bone marrow forms a clot at the lesion site which is an enriched environment for new tissue formation. With the subject's consent a cartilage biopsy will be taken (at least 150 mg) and about 80 ml venous blood withdrawn. This will be used for chondrocyte culture and cryopreservation in case a later BioCart™II implantation is required after failure of the microfracture procedure.
  Other Names: MF
  Arms: B

SUMMARY:
BioCart™II is a novel scaffold seeded with autologous chondrocytes to be used to repair cartilage lesions of the knee. This study is designed to compare the efficacy and safety of BioCart™II treatment compared to microfracture which is the classical method of treatment.

DETAILED DESCRIPTION:
Full thickness cartilage lesions are typically incapable of self repair, are a source of pain and morbidity and lead to early onset osteoarthritis. A classical method of treatment has been microfracture where holes are drilled in the subchondral bone to allow influx of bone marrow cells which fill and repair the lesion. The resulting repair has been reported to be mixed fibrocartilage which is recognized to be less efficient and durable than hyaline cartilage, the physiological material making up the joint. In autologous chondrocyte implantation, a sample of cartilage is removed from a non-weight bearing region of the joint and the cells are grown and expanded in culture and then returned to the knee to repair the damaged cartilage. For implantation with BioCart™II, the chondrocytes are grown in the presence of proprietary growth factors which maintain the chondrocytes in optimal condition for subsequent repair. For implantation, the cells are seeded on a completely human three dimensional spongelike scaffold which holds the cells in the correct topology to allow for a rapid repair of the damaged joint with true physiological cartilage. BioCart™II is user friendly for the surgeon and patient alike giving it an advantage over other methods for autologous chondrocyte implantation that are in clinical use.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 to 60 years
* Femoral condyle lesion (medial, lateral or trochlea)
* Single contained lesion
* Symptomatic (moderate to severe pain on VAS)
* Caused by trauma or OCD
* Depth of lesion up to 6 mm
* Size of lesion 1.5-7.5 cm2
* No general bone or cartilage pathology
* No limb mal-alignment (long leg standing X-ray)
* Mechanically stable knee
* Accompanying pathology menisectomy up to 50%
* Willing and able to comply with protocol and undergo vigorous rehabilitation
* Signed informed consent

Exclusion Criteria:

* Multiple cartilage lesions of the knee, other location than femoral condyle (medial, lateral or trochlear), deeper than 6 mm, smaller than 1.5cm2 or greater than 7.5cm2, mild symptoms, caused by reason other than trauma or OCD, unstable knee, accompanying pathology other than 50% menisectomy.
* Hyaluronic acid knee injections in the past 3 months,
* History of chronic bone or cartilage disorder, bilateral knee pain and/or cartilage lesion
* History of any neoplastic disease, or chemotherapy treatment
* Chronic steroid intake, chronic pain medication use for conditions other than the involved knee, use of blood thinners (during the past 10 days prior to enrollment)
* History of allergy or atopic disease, sensitivity to blood products
* Evidence of any significant systemic disease, known coagulopathies or acute injury that might compromise the patient's welfare
* Pregnant or lactating women
* Substance or alcohol abuse
* Microfracture to the affected knee within the previous 2 years
* Participation in concurrent trials
* Participation in previous trials within 3 months
* Malignancy
* Taking specific drugs for osteoarthritis, such as chondroitin sulfate, diacerein, n-glucosamine, piaseledine, or capsaicin within 2 weeks of the baseline visit
* Chronic use of anticoagulants
* Uncontrolled diabetes
* Active joint infection
* Other unstable cardiac and pulmonary disorder
* Liver enzymes (SGOT, SGPT, alkaline phosphatase) of more then two times the upper limit of normal or any other results that in the clinical investigator's mind is important clinically
* Clinical and/or radiographic disease in the indexed affected joint that includes:
* Osteoarthritis or avascular necrosis
* Rheumatoid arthritis or a history of septic or reactive arthritis
* Gout or a history of gout or pseudogout in the affected knee
* Osteochondritis dissecans of the knee with significant bone loss
* Bipolar articular cartilage involvement (or kissing lesions) of the ipsilateral compartment (i.e >than ICRS grade 2 on the opposing articular surface)
* Associated damage to the underlying subchondral bone requiring an osteochondral graft
* History of secondary arthropathies (i.e. sickle cell disease, Hemochromatosis, or autoimmune disease)
* Receiving prescription pain medication other than NSAIDs or acetaminophen for conditions unrelated to the index knee conditions
* BMI >40 kg/m2
* Unable to undergo MRI
* Any reasons making the patient a poor candidate in the eyes of the investigator

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-05; Primary Completion 2012-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Improvement in the Lysholm joint function score of subjects in the BioCart™II study group compared with the MF study group | 12 months with optional follow up to 5 years

SECONDARY OUTCOMES:
Improvement in clinical function post implantation/surgery compared to baseline in the study group and compared with the control group, of the following: | 12 months with optional follow up to 5 years
IKDC knee score | 12 months with optional follow up to 5 years
KOOS questionnaire | 12 months with optional follow up to 5 years
ICRS functional status | 12 months with optional follow up to 5 years
VAS pain score | 12 months with optional follow up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Avner Yayon, PhD MD, Study Director — ProChon Biotech Ltd
Locations (8):
- United States (5):
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - Southeastern Orthopedic Center, Savannah, Georgia
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Mount Sinai Medical Center, New York, New York
  - University Orthopedics Center, Altoona, Pennsylvania
- Israel (3):
  - Sheba Medical Center Tel Hashomer, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Assaf Harofeh Medical Center, Ẕerifin

REFERENCES:
- [Background] Nehrer S, Chiari C, Domayer S, Barkay H, Yayon A. Results of chondrocyte implantation with a fibrin-hyaluronan matrix: a preliminary study. Clin Orthop Relat Res. 2008 Aug;466(8):1849-55. doi: 10.1007/s11999-008-0322-4. Epub 2008 Jun 5. PMID 18528742
- [Background] Domayer SE, Welsch GH, Nehrer S, Chiari C, Dorotka R, Szomolanyi P, Mamisch TC, Yayon A, Trattnig S. T2 mapping and dGEMRIC after autologous chondrocyte implantation with a fibrin-based scaffold in the knee: preliminary results. Eur J Radiol. 2010 Mar;73(3):636-42. doi: 10.1016/j.ejrad.2008.12.006. Epub 2009 Jan 20. PMID 19157740